CLINICAL TRIAL: NCT04390438
Title: Efficacy of High and Low Intensity Percutaneous Electrolysis for the Treatment of Myofascial Pain Syndrome: A Pilot Study
Brief Title: Efficacy of High and Low Intensity Percutaneous Electrolysis for the Treatment of Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 50997093
Record Dates: First submitted 2020-04-30; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-04

CONDITIONS: Knee Pain Chronic; Muscle Pain
Keywords: Patellofemoral pain syndrome; Electrolysis; Myofascial Pain Syndromes; Acupuncture
MeSH Terms: conditions — Myalgia; Patellofemoral Pain Syndrome; Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Randomized Clinical trial with 3 parallel groups; 2 experimental groups and 1 control group
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Intensity short time percutaneous electrolysis (Experimental): Application of a 0,66uA galvanic current in the active TrP through a needle during 10 seconds. During the 20 seconds left necessary to blind the patient and the examiner, the needle was inside but with no electrical current
  Interventions: Procedure: Percutaneous Electrolysis
- Low-Intensity long time percutaneous electrolysis (Experimental): Application of a 0,22uA galvanic current in the active TrP through a needle during 30 seconds
  Interventions: Procedure: Percutaneous Electrolysis
- Dry needling (Active Comparator): One acupuncture needle was placed in the active TrP to produce a local twitch response during 30 seconds
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Percutaneous Electrolysis — Needle emplacement with a galvanic electrical current
  Arms: High-Intensity short time percutaneous electrolysis; Low-Intensity long time percutaneous electrolysis
Procedure: Dry needling — Needle emplacement without electrical current nor substance
  Arms: Dry needling

SUMMARY:
Muscle pain is frequently attributed to myofascial pain syndrome (MPS) in which myofascial trigger points (MTrP) are a characteristic feature. Dry needling is a frequent clinical practice to manage MPS but few evidence is published about percutaneous electrolysis effects for the treatment of MPS.

This is a randomized clinical trial with 3 parallel groups: 1) High intensity-short time percutaneous electrolysis; 2) Low intensity-long time percutaneous electrolysis; 3) dry needling control group.

DETAILED DESCRIPTION:
The current study aimed to evaluate changes in rectus femurs active trigger points and patellar tendon pain pressure thresholds and subjective anterior knee pain perception after application of two percutaneous electrolysis methods using a same charge (high intensity and low intensity) compared to a dry needling group in patients with patellofemoral pain syndrome (PFPS)

Fifteen patients diagnosed with unilateral PFPS were divided in two experimental groups (high intensity percutaneous electrolysis and low intensity percutaneous electrolysis) and one active control group (dry needling. The duration of the study was 7 days with only one intervention. Pain pressure thresholds were assessed using an algometer before the intervention, immediately after the intervention and after 7 days and a Visual Analogue Scale was used before the treatment and after 7 days to rate the subjective anterior knee pain perception. Also a VAS was used to rate the pain perception during the intervention

ELIGIBILITY:
Inclusion Criteria:

* Athletes with knee pain
* Presence of at least one active Trigger point

Exclusion Criteria:

* Farmacologic treatment
* Surgery or traumas
* Skin alterations or infections
* Prior 6 weeks DN nor PT treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold (Trigger Point) | 7 days
  Algometry (Wagner analogical algometer)
Pressure Pain Threshold (Patellar Tendon) | 7 days
  Algometry (Wagner analogical algometer)

SECONDARY OUTCOMES:
Subjective pain perception | 7 days
  Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Valera-Calero, PT, Msc, Principal Investigator — Camilo Jose Cela University; Alberto Sanchez-Mayoral-Martín, PT, Study Director — Free professional practice
Locations (1):
- Camilo Jose Cela University, Villanueva de la Cañada, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No